CLINICAL TRIAL: NCT01795625
Title: A Multi-centre, Open Clinical Evaluation to Determine Professional Clinical Accuracy Comparing the OneTouch® Verio™Pro+ Blood Glucose Results With the YSI 2300 Analyzer.
Brief Title: OneTouch® Verio™Pro+ Blood Glucose Monitoring System Clinical Accuracy Study in China
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Medical, China (Industry)
Responsible Party: Sponsor
Other Study IDs: LFS-201201
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Blood Glucose Measurement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The evaluation will determine professional clinical accuracy comparing the OneTouch® Verio™Pro+ blood glucose results with the YSI 2300 analyzer. "Professional Clinical Accuracy" is defined as accuracy of the system when used by a trained healthcare professional.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age.
* Subject has been diagnosed with diabetes mellitus (type 1 or type 2 diabetes)
* Subject agrees to sign two (2) copies each of the Subject Informed Consent Form and to follow the procedures of the study.
* Subject agrees to allow the HCP to perform finger stick for blood glucose test by the meter and the YSI instrument. Up to one retry of finger stick will be needed in the event of insufficient blood collected or test failure.
* Subject agrees to allow the HCP to perform venous puncture for blood glucose test by the meter and the YSI instrument, and for haematocrit (HCT) test. Up to one retry of venous puncture will be needed in the event of insufficient blood collected or test failure.
* Subject agrees to provide demographic and medical history information and give access to medical records where appropriate.

Exclusion Criteria:

* Subject is currently working for, has previously worked for, or has an immediate family member working for a company manufacturing and/or marketing blood glucose monitoring products.
* Subject has already participated in this study.
* Subject is known pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of at least 240 diabetic subjects (type 1 or type 2) study-wide at two clinical sites.
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2012-08-31 (Actual); Primary Completion 2012-10-31 (Actual); Study Completion 2012-10-31 (Actual)

PRIMARY OUTCOMES:
• Obtain professional clinical accuracy data for the OneTouch® Verio™Pro+ blood glucose monitoring meter in comparison with a standard laboratory reference (YSI 2300 glucose analyzer) using a capillary blood sample and a venous sample | 56days
  August 20,2012~October 14,2012

CONTACTS AND LOCATIONS:
Overall Officials: Yongde Peng, Professor, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Fengling Chen, Professor, Principal Investigator — Shanghai Jiaotong University, medical school affiliated Third People's Hospital
Locations (2):
- China (2):
  - Shanghai First People's Hospital, Shanghai
  - Shanghai Jiaotong University, medical school affiliated Third People's Hospital, Shanghai